CLINICAL TRIAL: NCT01542866
Title: A 16 Week Evaluation of the Novartis Health Management Tool in Assessing Self-test Visual Function in Patients With AMD Treated With Ranibizumab
Brief Title: A 16 Week Evaluation of the Novartis Health Management Tool (HMT) in Age Related Macular Degeneration (AMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Carematix, VAS (Vital Art and Science) (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRFB002A2407
Record Dates: First submitted 2011-07-01; First posted 2012-03-02 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Age Related Macular Degeneration (AMD)
Keywords: ranibizumab; Age related Macular Degeneration; AMD; Health Management Tool; HMT; Best Corrected Visual Acuity; Investigator's Clinical Judgement of Change; Choroidal Neovascularization; Central Retinal Subfield Thickness; visual function self test
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Monitoring Test (Experimental): Health management tool (HMT) for measuring vision impairment
  Interventions: Other: Health Management Tool (HMT)

INTERVENTIONS:
Other: Health Management Tool (HMT) — Mobile computing platform (ie HMT) which allows subjects to perform home monitoring tests

SUMMARY:
This is a prospective pilot study to evaluate the usability and applicability of a self monitoring test of visual function with the handheld Health Management Tool (HMT) to remotely monitor neovascular Age Related Macular Degeneration (AMD) to detect a potential change in disease status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CNV secondary to AMD and not other causes in at least one eye identified by the investigator to be eligible for ranibizumab treatment
* Patients with a BCVA letter score in the study eye is 24 or better using an ETDRS chart measured at 4 meters distance

Exclusion Criteria:

* Patients with any concurrent ocular condition that may result in visual loss during the study
* Patients with past (within the prior 6 months) or current use of, or likely need for, systemic medications that are known to be toxic to the lens, retina, or optic nerve
* Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-01-11 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2011-11-30 (Actual)

PRIMARY OUTCOMES:
Threshold value of handheld Health Management Tool (HMT) for choroidal neovascular AMD diagnosis at baseline | 16 weeks
Identification of clinically relevant worsening of visual function in the home self testing mVT scores | baseline to 16 weeks

SECONDARY OUTCOMES:
Correlation of the handheld Health Management Tool (HMT) home self testing on the days of site visits and the mVT assessments performed during the site visits for absolute values | after 16 weeks
Correlation between the home deterioration signal and the monthly change in the handheld Health Management Tool (HMT) assessments performed during the site visits | after 16 weeks
Patient compliance and reliability of performing the home self testing using the handheld Health Management Tool (HMT) | after 16 weeks
Correlation between absolute values of the handheld Health Management Tool (HMT) and BCVA/ central retinal subfield thickness (CRST) | 16 weeks
Correlation of the monthly changes in handheld Health Management Tool(HMT)to those of BCVA / OCT / Clinical examination | after 16 weeks
Correlation of diagnosis of choroidal neovascular AMD with BCVA/ central retinal subfield thickness | baseline
  The disease diagnoses at baseline will be correlated to values of BCVA and CRST at baseline
Correlation of monthly changes observed with thein the investigator judgment (CJ-C) to BCVA / OCT / Clinical examination | baseline to 16 weeks
  Monthly changes in BCVA /OCT and clinical examination will be compared to clinical relevant changes as judged by the investigator on the CJC.
Patient compliance with the signs and symptom questionnaire | baseline to 16 weeks
  The percentage of completed assessments of the signs & symptoms questionnaire on the HMT will be provided
Patient satisfaction regarding the use of the HMT | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (23):
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Williamsburg, Michigan
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Toms River, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Slingerlands, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, West Mifflin, Pennsylvania
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, San Antonio, Texas